CLINICAL TRIAL: NCT02808221
Title: Readmission in the Case of Patients With Heart Failure
Acronym: PRADO-IC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6361
Record Dates: First submitted 2016-04-12; First posted 2016-06-21 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure
Keywords: Heart failure; heart disease; left ventricular
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) is a serious chronic disease with frequent readmissions, some of which can be prevented by early action. The management of HF is complex: long, often difficult and costly. In France, nearly one million people suffer from HF and 120,000 new cases are diagnosed every year. With the aging population, this number will continue to evolve and become a real public health problem. Within 10 to 20 years ahead, WHO projects that heart failure in either the 3 most common diseases in industrialized countries.

Investigators goals are to make an inventory of PRADO-IC project in terms of its effectiveness on readmission of patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient readmitted for heart failure

Exclusion Criteria:

* Population whose age is less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The cost of re-hospitalization in the case of patients with heart failure reach | during 2015

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ANDRES, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Médecine Interne, diabète et maladies métaboliques - Médicale B, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No